CLINICAL TRIAL: NCT02127385
Title: The Type of Hepatoglobin in IUGR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0001-14
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Haptoglobin Type

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Blood test for H-p genotype
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IUGR

SUMMARY:
Intra Uterine Growth Restriction is associated with increased oxidative stress. Haptoglobin (Hp) is an abundant plasma glycoprotein produced in the liver. The function of Hp is as anti oxidant agent, it binds free hemoglobin (Hb) released from red blood cells to decrease oxidative tissue damage. There are 3 differenet genotype of haptoglobin Hp 1-1 Hp 1-2 and Hp 2-2 with different anti oxidant properties and different prevalence ( Hp 1-1, Hp 1-2 and Hp 2-2approximately 16%, 48% and 36% respectively) . we hypotheise that IUGR will be more common and severe in the Hp 2-2 genotype with the less anti oxidant properties.

ELIGIBILITY:
Inclusion Criteria: Pregnancies complicated with IUGR -

Exclusion Criteria: NOT INTERESTED DO PARTICIPATE

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients adimitted with IUGR
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
type of haptoglobin | 10 weeks
  severity of iugr

CONTACTS AND LOCATIONS:
Overall Officials: RON BELOOSESKY, M.D, Principal Investigator — HILLEL YAFFE MEDICAL CENTER- TECHNION